CLINICAL TRIAL: NCT05980793
Title: Denervation for Osteoarthritis in the PIP-joint Efficacy Study (DOPS), a Randomized Controlled Trial
Brief Title: Denervation for Osteoarthritis in the PIP-joint Efficacy Study (DOPS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Elin Swärd, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DOPS
Record Dates: First submitted 2023-06-29; First posted 2023-08-08 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis Finger; Surgery
MeSH Terms: interventions — Patient Education as Topic; Exercise

STUDY DESIGN:
Intervention Model Description: A parallel group, two-arm, randomized, controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Data analysts will be masked for treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical treatment (Active Comparator): PIP joint denervation is performed through a volar approach.
  Interventions: Procedure: PIP joint denervation
- Non-surgical treatment (Active Comparator): An education and exercise program.
  Interventions: Procedure: Patient education plus exercise

INTERVENTIONS:
Procedure: PIP joint denervation — Surgical denervation of the PIP joint
  Arms: Surgical treatment
Procedure: Patient education plus exercise — An education plus exercise program
  Arms: Non-surgical treatment

SUMMARY:
The goal of this clinical trial is to compare the effects of a surgical and a non-surgical treatment method in patients with osteoarthritis in the proximal interphalangeal (PIP) joint. The main questions it aims to answer are:

* Are the treatments effective?
* Is the surgical treatment more effective than the non-surgical treatment? Participants will receive surgical treatment (PIP joint denervation) or non surgical treatment (patient education plus exercise).

Researchers will compare the non-surgical and surgical groups to see if pain, patient-reported function, quality of life, movement and grip strength differs between the groups.

DETAILED DESCRIPTION:
This is a parallel group, two-arm, randomized, controlled trial comparing the effects of surgical denevation to patient education plus exercise in patients with symptomatic PIP joint osteoarthritis.

The research questions are:

1. Does any of the treatments denervation of the PIP-joint and patient education plus exercise decrease pain, improve patient-reported outcomes, grip strength and range of motion (ROM) in PIP-joint osteoarthritis?
2. Does denervation of the PIP-joint decrease pain, and improve patient-reported outcomes grip strength and ROM more effectively than patient education plus exercise for PIP-joint osteoarthritis?

Participants will be randomly assigned (1:1) to receive surgical denervation of the PIP-joint or education plus exercise. A block randomization scheme with a fixed block size of 10 will be used. Patients will be stratified according to gender. Sealed opaque envelopes will be used and data analysts will be masked for treatment allocation.

Assesments will be made at inclusion, and after 3, 6 and 12 months. The studys primary enpoint is 12 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Chronic symptomatic osteoarthritis in the PIP-joint.
* Radiological signs of osteoarthritis on posteroanterior and lateral radiographs assessed by the Kellgren-Lawrence classification (grade II-IV) (Kellgren & Lawrence, 1957).
* Clinical signs of PIP-joint arthritis.

Exclusion Criteria:

* Inflammatory arthritis.
* Ongoing infection in the hand.
* Inability to co-operate with the follow-up protocol.
* Intra-articular glucocorticoid, PRP or Hyaluronic acid injections in the affected joint less than 3 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2028-07-15 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
Pain on load (change baseline to -12 months) | 0-12 months
  Pain (Numerical Rating Scale, 0-100 points, 100 is a worse outcome)

SECONDARY OUTCOMES:
Pain at rest (change baseline to -3, -6, -12 months) | 0-12 months
  Pain (Numerical Rating Scale, 0-100 points, 100 is a worse outcome)
HQ8 (8-item patient questionnaire) change baseline to -3, -6, 12 months | 0-12 months
  A questionnaire used by Swedish Healthcare Quality Registry for hand surgery (HAKIR), 0-100 points, 100 is a worse outcome.
PRWHE (Patient Rated Wrist/Hand Evaluation) change baseline to -3, 6, 12 months | 0-12 months
  A questionnaire that measures hand/wrist function (0-100 points, 100 is a worse outcome)
EQ5D-5L change baseline to -3, -6, -12 months | 0-12 months
  A questionnaire that measures quality of life (0-1 point, 0 is a worse outcome).
Objective function change baseline to -3, -6, -12 months | 0-12 months
  Range of motion (goniometer with 5 degrees interval)
Objective function change baseline to -3, -6, -12 months | 0-12 months
  grip strength (hydraulic hand dynamometer, kilograms)
Complications | 0-12 months
  2PD (Two point discrimination, 0-15mm, 15 indicating a worse outcome)
Complications | 0-12 months
  Mini Sollerman (0-12 points, 12 indicating a better outcome)
Complications | 0-12 months
  Infection (clinical evaluation, positive cultures, need for antibiotics)
Additional treatment | 0-12 months
  Need for further surgery/treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elin Sward, MD, PhD, Principal Investigator — Department of Hand Surgery Sodersjukhuset and Karolinska Institutet
Locations (1):
- Department of Hand Surgery, Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sward EM, Beckman J, Tabaroj F, Wilcke MK. Efficacy of denervation for osteoarthritis in the proximal interphalangeal joint (DOP): protocol of a randomized controlled trial. Trials. 2024 Aug 22;25(1):553. doi: 10.1186/s13063-024-08399-w. PMID 39169395